CLINICAL TRIAL: NCT01569477
Title: Striving to Quit: Wisconsin Tobacco Quit Line Tobacco Cessation Research
Brief Title: Striving to Quit-Wisconsin Tobacco Quit Line
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit participants
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0198
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Smoking Cessation; Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment incentives (Experimental): Incentives for biochemical verification visits, treatment engagement, and abstinence
  Interventions: Behavioral: Incentives for abstinence and treatment engagement
- Attendance incentive (Active Comparator): Incentives for only attending the biochemical verification visits
  Interventions: Behavioral: Attendance incentive

INTERVENTIONS:
Behavioral: Incentives for abstinence and treatment engagement — Treatment incentives - incentives for biochemical verification visits, treatment engagement and abstinence
  Arms: Treatment incentives
Behavioral: Attendance incentive — Attendance Incentives - incentives for only attending the biochemical verification visits
  Arms: Attendance incentive

SUMMARY:
This study is designed to test the hypotheses that incentives can increase both participation in smoking cessation treatment and resulting cessation rates when they are offered to Medicaid BadgerCare Plus members.

DETAILED DESCRIPTION:
Aim 1: To determine the extent to which contingent financial "treatment incentives" (i.e., incentives for biochemical verification visits, treatment engagement, and abstinence) versus "attendance incentives" (i.e., incentives for only attending the biochemical verification visits), increase rates of smoking cessation . Participants will be BadgerCare Plus tobacco users who enroll in Wisconsin Tobacco Quit Line (WTQL) services.

Aim 2: To determine the extent to which treatment incentives vs. attendance incentives increase rates of engagement in smoking cessation treatment through the WTQL when offered to BadgerCare Plus members who smoke.

Aim 3: To determine the cost-effectiveness of the smoking cessation program when paired with treatment incentives and when paired with attendance incentives.

Aim 4: To identify moderating and mediational effects regarding the clinical benefit of incentivized smoking treatment

Aim 5: To determine the reach of an incentivized smoking cessation treatment that depends upon primary care clinic staff, a fax-to-quit referral mechanism and a state quit line.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in Wisconsin Medicaid (BadgerCare Plus)
* resides in study area (one of 25 counties)
* member of participating HMOs
* 18 or older
* English speaking
* has smoked daily (at least 5 cigarettes each day) over the last week
* willingness to attend visits at his/her PCC (primary care clinic) every 6 months (3 times over a 12 month period), provide urine samples, and complete follow-up phone calls
* willingness to inform the WTQL as to any change in address, phone number, clinic attended, or health plan.

Exclusion Criteria:

* not enrolled in Wisconsin Medicaid (BadgerCare Plus)
* not reside in study area
* not a member participating HMOs
* less than 18 years of age
* not English speaking
* does not smoke daily (at least 5 cigarettes each day) over the last week
* not willing to attend visits at his/her PCC (primary care clinic) every 6 months (3 times over a 12 month period), provide urine samples, and complete follow-up phone calls.
* not willing to inform the WTQL as to any change in address, phone number, clinic attended, or health plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Abstinence from smoking | Measured 6 months after enrollment at follow-up assessment
  The data will be the biochemically confirmed reports of abstinence for the past 7 days (i.e., 7-day point-prevalence abstinence)

SECONDARY OUTCOMES:
Engagement in treatment | Measured 12 months after enrollment at follow-up assessment
  The primary analyses will compare number of calls completed
Cost-effectiveness | Measured 12 months after enrollment
  The primary analysis will contrast the incremental costs of the treatment vs. attendance conditions by computing the Incremental Cost-Effectiveness Ratio (ICER) with regard to attaining 6-month abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Baker, PhD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: Yes